CLINICAL TRIAL: NCT02588092
Title: A Phase 1, Open-label, Dose-escalation, Multicenter Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Activity of ADCT 301 in Patients With Relapsed or Refractory CD25-positive Acute Myeloid Leukemia (AML) or CD25-positive Acute Lymphoblastic Leukemia
Brief Title: Study of ADCT-301 in Patients With Relapsed/Refractory CD25-positive Acute Myeloid Leukemia (AML) or CD25-positive Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-301-002
Record Dates: First submitted 2015-08-13; First posted 2015-10-27 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Camidanlumab tesirine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: ADCT-301 (dose escalation) (Experimental): Weekly administration - Participants will receive an IV infusion of ADCT-301, on Days 1, 8, and 15 of each 3-week (21-day) cycle.
  3-week administration - Participants will receive an IV infusion of ADCT-301, on Day 1 of each 3-week (21-day) cycle.
  The dose escalation will be conducted according to a 3+3 design.
  Interventions: Drug: ADCT-301
- Part 2: ADCT-301 (dose expansion) (Experimental): Participants will be assigned to receive the recommended dose and/or schedule of ADCT-301 as determined by the Dose Escalation Steering Committee.
  Interventions: Drug: ADCT-301

INTERVENTIONS:
Drug: ADCT-301 — Intravenous infusion
  Other Names: Camidanlumab tesirine

SUMMARY:
This study evaluates ADCT-301 in participants with Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL). Participants will participate in a dose-escalation phase (Part 1) and receive ADCT-301 either weekly or once every 3 weeks.

In Part 2 of the study, participants will receive a recommended dose of ADCT-301 as determined by a Dose Escalation Steering Committee.

DETAILED DESCRIPTION:
This is a Phase 1 study with ADCT-301 to evaluate the safety, tolerability and pharmacokinetics of ADCT-301 in participants with Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL).

ADCT-301 is a human monoclonal antibody attached via a cleavable linker to a pyrrolobenzodiazepine (PBD) warhead which, when internalized by antigen expressing cells, covalently cross links deoxyribonucleic acid (DNA) preventing replication.

The study will be conducted in 2 parts: In Part 1 (dose escalation) participants will either be on weekly administration or every 3-week administration. Participants on weekly administration will receive an infusion of ADCT-301 on Days 1, 8, and 15 of each 3 week treatment cycle. Participants on 3-week administration will receive an infusion of ADCT-301 on Day 1, every 3 weeks. Dose escalation will continue until the maximum tolerated dose (MTD) is determined.

In Part 2 (expansion), participants will be assigned to receive a recommended dose and/or schedule of ADCT-301 as determined by a Dose Escalation Steering Committee.

For each participant, the study will include a screening period (up to 28 days), a treatment period, and a follow-up period to assess disease progression and survival for up to 12 months after the last dose of study drug. The total study duration will be dependent on overall participant tolerability to the study drug and response to treatment. It is anticipated that the entire study (Parts 1 and 2) will enroll a maximum of 80 participants and could last approximately 3 years from first participant treated to last participant completed.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD25-positive AML [per World Health Organization (WHO)].
* Relapsed or refractory CD25-positive ALL [per World Health Organization (WHO)].
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Creatinine ≤1.5mg/dL.
* Serum/plasma alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤2 times the upper limit of normal (ULN); ≤5 times ULN if there is liver or bone involvement.
* Total serum/plasma bilirubin ≤1.5 times the upper limit of normal.
* Women of childbearing potential must have a negative urine or serum beta-human chorionic gonadotropin pregnancy test within 7 days prior to Day 1.
* Women of childbearing potential must agree to use a highly effective method of contraception. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception.
* White Blood Cell Count value of <15,000 cells/μL prior to Cycle 1 Day 1.

Exclusion Criteria:

* Participants who have an option for any treatment with proven clinical benefit for CD25-positive AML or CD25-positive ALL at current state of disease.
* Known active central nervous system (CNS) leukemia, defined as morphologic evidence of leukemic blasts in the cerebrospinal fluid (CSF), use of CNS directed intrathecal treatment for active disease within 28 days prior to Screening, or symptomatic CNS leukemia (i.e., cranial nerve palsies or other significant neurologic dysfunction) within 28 days prior to Screening.
* Active graft versus host disease.
* Autologous or allogenic transplant within the 60 days prior to Screening.
* Known history of immunogenicity or hypersensitivity to a CD25 antibody.
* Known history of positive serum human anti-drug antibodies (ADA), or known allergy to any component of ADCT-301.
* Active autoimmune disease; other CNS autoimmune disease. Known seropositive for human immunodeficiency (HIV) virus, hepatitis B surface antigen (HbsAg), or antibody to hepatitis C virus (anti-HCV) with confirmatory testing and requiring anti-viral therapy.
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis syndrome.
* Pregnant or breastfeeding women.
* Significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure >115 mm Hg), unstable angina, congestive heart failure (greater than New York Heart Association class II), severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty, myocardial infarction within 6 months prior to Screening, or uncontrolled atrial or ventricular cardiac arrhythmias.
* Use of any other experimental medication(s) within 14 days or 5 half-lives but in no case < 14 days prior to the start of the study treatment on Cycle 1, Day 1.
* Major surgery, chemotherapy, systemic therapy (excluding hydroxyurea, steroids, and any targeted small molecules or biologics), or radiotherapy, or biotherapy targeted therapies within 14 days or 5 half-lives (whichever is shorter) prior to Cycle 1, Day 1 treatment, except if approved by the Sponsor.
* Failure to recover (to CTCAE Version 4.0 Grade 0 or Grade 1) from acute non hematologic toxicity (except all grades of alopecia or Grade 2 or lower neuropathy), due to previous therapy, prior to Screening.
* Isolated extramedullary relapse (i.e., testicular, CNS).
* Congenital long QT syndrome or a corrected QT interval (QTc) ≥450 ms at Screening (unless secondary to pacemaker or bundle branch block).
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy.
* Any other significant medical illness, abnormality, or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Goldberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Greenville Health System, Institute for Translational Oncology Research, Greenville, South Carolina
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital/ Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg AD, Atallah E, Rizzieri D, Walter RB, Chung KY, Spira A, Stock W, Tallman MS, Cruz HG, Boni J, Havenith KEG, Chao G, Feingold JM, Wuerthner J, Solh M. Camidanlumab tesirine, an antibody-drug conjugate, in relapsed/refractory CD25-positive acute myeloid leukemia or acute lymphoblastic leukemia: A phase I study. Leuk Res. 2020 Aug;95:106385. doi: 10.1016/j.leukres.2020.106385. Epub 2020 Jun 7. PMID 32521310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 sites in the United States between 01 February 2016 and 29 August 2018.
Groups:
- Cohort 1: 3 μg/kg Q3W: Participants received 3 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 2: 6 μg/kg Q3W: Participants received 6 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 3: 12 μg/kg Q3W: Participants received 12 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 4: 22 μg/kg Q3W: Participants received 22 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 5: 32 μg/kg Q3W: Participants received 32 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle.
- Cohort 6: 52 μg/kg Q3W: Participants received 52 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 7: 72 μg/kg Q3W: Participants received 72 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 8: 92 μg/kg Q3W: Participants received 92 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Cohort 9: 30 μg/kg QW: Participants received 30 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Days 1, 8 and 15 (once weekly [QW]) of each 3-week (21 day) cycle.
- Cohort 10: 37.5 μg/kg QW: Participants received 37.5 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Days 1, 8 and 15 (once weekly [QW]) of each 3-week (21 day) cycle.
Period: Overall Study
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Started | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3
Not completed — Death | 4 | 3 | 3 | 3 | 2 | 2 | 2 | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Started Another Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 5: 32 μg/kg Q3W: Participants received 32 μg/kg ADCT-301 formulation, intravenous infusion for 1 hour, on Day 1 of each 3-week (21-day) cycle (Q3W).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 2 | 12
  >=65 years | 2 | 3 | 1 | 1 | 3 | 2 | 3 | 2 | 5 | 1 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (11.09) | 72.3 (4.73) | 51.0 (17.78) | 51.7 (26.27) | 69.3 (2.89) | 67.0 (13.00) | 75.7 (5.69) | 56.5 (18.43) | 71.0 (10.77) | 63.3 (10.02) | 64.9 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 10
  Male | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4 | 6 | 3 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 35
Height [Mean (Standard Deviation); unit: cm] — Population: Height data was not collected for one participant because of complications during the collection of baseline measurements.
  cm
    number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 34
    (all) | 169.40 (10.641) | 179.27 (15.255) | 183.20 (9.354) | 170.00 (4.359) | 176.33 (4.856) | 165.50 (18.007) | 168.57 (6.562) | 169.38 (11.762) | 169.52 (12.478) | 177.22 (3.586) | 172.44 (10.774)
Weight [Mean (Standard Deviation); unit: kg] | 94.98 (24.758) | 99.30 (12.644) | 73.50 (7.988) | 72.20 (11.722) | 105.67 (24.509) | 71.63 (15.053) | 71.67 (11.395) | 79.45 (17.436) | 74.10 (5.686) | 75.23 (5.200) | 81.43 (17.597)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI could not be analyzed for one participant because height data was not collected.
  kg/m^2
    number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 34
    (all) | 29.37 (3.100) | 31.09 (4.209) | 21.94 (2.469) | 24.89 (3.002) | 33.86 (7.003) | 25.98 (1.259) | 25.52 (6.243) | 27.47 (3.759) | 26.03 (3.607) | 23.94 (0.934) | 26.94 (4.656)
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG performance status is graded from 0 to 5:
  0: Fully active, able to carry on all predisease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
  Participants
    0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    1 | 3 | 3 | 2 | 2 | 3 | 2 | 2 | 3 | 5 | 2 | 27
    2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLT)
Description: A DLT is defined as any of the following events, except those that are clearly due to underlying disease or extraneous causes:
  A hematologic DLT is defined as:
  - Grade 3 or higher event of neutropenia or thrombocytopenia, or a Grade 4 anemia, with a hypocellular bone marrow lasting for 6 weeks or more after the start of a cycle, in the absence of residual leukemia (i.e., with <5% blasts). In case of a normocellular bone marrow with <5% blasts, 8 weeks with ≥Grade 3 pancytopenia will be considered a DLT.
  A non-hematologic DLT is defined as:
  * Grade 4 tumor lysis syndrome.
  * Grade 3 or higher AE (including nausea, vomiting, diarrhea, and electrolyte imbalances lasting more than 48 hours despite optimal therapy; excluding all grades of alopecia).
  * CTCAE Grade 3 or higher hypersensitivity reaction (regardless of premedication).
  * CTCAE Grade 3 or higher skin ulceration.
  * Peripheral sensory or motor neuropathy ≥ Grade 2.
Time Frame: Day 1 to Day 21 (Cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Recommended Dose of ADCT-301 for Part 2
Description: The recommended dose was to be established by the dose escalation steering committee and based on safety findings during part 1 of the study.
Time Frame: Day 1 to Day 21 (Cycle 1)
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Groups:
- Part 1: ADCT-301 Dose Escalation: Weekly administration: Participants received an IV infusion of ADCT-301, on Days 1, 8, and 15 of each 3-week (21-day) cycle.
  3-week administration: Participants received an IV infusion of ADCT-301, on Day 1 of each 3-week (21-day) cycle.
  The dose escalation was conducted according to a 3+3 design.
Arm/Group | Part 1: ADCT-301 Dose Escalation
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is defined as any adverse event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug.
Time Frame: Day 1 to a maximum of 24 weeks (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3
Participants | 4 | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3

4. Primary Outcome: Number of Participants Reporting One or More Treatment Emergent Serious Adverse Event (SAE)
Description: An SAE is defined as any event that results in death, is immediately life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. Hospitalization for elective procedures or for protocol compliance is not considered an SAE.
Time Frame: Day 1 to a maximum of 24 weeks (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3
Participants | 2 | 1 | 2 | 3 | 1 | 2 | 2 | 2 | 5 | 3

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined among responders (complete response [CR], CR with incomplete blood count recover [CRi], or partial response [PR]) as the time from the earliest date of first response until the first date of either disease progression or death due to any cause. A summary of antitumor activity was not conducted due to a limited number of responders.
  CR:
  * Bone marrow differential showing ≤5% blast cells.
  * Absolute neutrophil count (ANC) ≥1.0 x 10^9/L and platelet count ≥100 x 10^9/L.
  * Absence of extramedullary disease.
  * Participant is independent of red blood cell transfusions.
  CRi is defined as achieving all CR criteria except that values for ANC may be <1.0 x 10^9/L and/or values for platelets may be <100 x 10^9/L.
  PR:
  * ANC ≥1.0 x 10^9/L and platelet count ≥100 x 10^9/L.
  * Bone marrow differential showing a ≥50% decrease from baseline in the percentage of bone marrow blast cells to a level >5% and ≤25%, or bone marrow differential showing <5% blast cells.
Time Frame: Screening, Day 19 visit (+/- 3 days) of Cycle 2 and each subsequent cycle up to 12 months after the last dose of study drug (1 cycle = 21 days)
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of CR, CRi, or PR at the time each participant discontinues treatment with ADCT-301. A summary of antitumor activity was not conducted due to a limited number of responders.
Time Frame: as for outcome 5
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of study drug treatment until the date of death due to any cause. A summary of antitumor activity was not conducted due to a limited number of responders.
Time Frame: as for outcome 5
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose of study drug until the first date of either disease progression or death due to any cause. A summary of antitumor activity was not conducted due to a limited number of responders.
Time Frame: as for outcome 5
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of ADCT-301 for the Q3W Dosing Schedule
Description: Cmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohorts.
Time Frame: Before infusion, end of infusion, 1, 3, 6, 24, 48, and 96 hours after infusion, and on Days 8 and 19 of Cycle 1 and 2 (1 cycle = 21 days)
Population: Only participants with evaluable pharmacokinetic results were included in the analysis. Where data is not presented, the pharmacokinetic profiles were nonmeasurable or short-lived in duration; therefore, no analysis could be performed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 2 | 1 | 3 | 3 | 3 | 3 | 4
μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  | 181 (348) | 165 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 186 (117) | 514 (127) | 920 (71.2) | 877 (35.4) | 949 (63.8)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 2 | 2 | 3
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  | 79.2 (0.268) |  | 589 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 405 (383) | 284 (102) | 1182 (167) | 710 (41.6)
  Total Ab of ADCT-301: Cycle 1 |  | 278 (355) | 177 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 233 (93.8) | 715 (139) | 960 (82.5) | 1013 (34.4) | 1196 (69.3)
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3 | 2 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  | 91.4 (17.0) |  | 272 (236) | 517 (330) | 333 (121) | 1406 (199) | 910 (41.0)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  SG3199 Free Warhead of ADCT-301: Cycle 1 |  |  |  |  |  | 0.0210 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0140 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0280 (54.3)
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  SG3199 Free Warhead of ADCT-301: Cycle 2 |  |  |  |  |  | 0.0140 (29.7) |  | 0.0170 (NA) — Standard deviation could not be determined as only one participant had evaluable data.

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of ADCT-301 for the QW Dosing Schedule
Description: Cmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: Before infusion, end of infusion, 5, 24, 48, and 96 hours after infusion on days 1 and 8, and before and after infusion on Day 15 of Cycle 1 and 2 (1 cycle = 21 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 5 | 2
μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1 | 377 (67.0) | 355 (39.4)
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2 | 350 (32.8) | 13200 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1 Week 1 | 435 (63.5) | 504 (22.2)
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  Total Ab of ADCT-301: Cycle 1 Week 2 | 416 (33.8) | 15100 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Reach the Maximum Observed Serum Concentration (Tmax) for ADCT-301 for the Q3W Dosing Schedule
Description: Tmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 2 | 1 | 3 | 3 | 3 | 3 | 4
days
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  | 0.162 (34.6) | 0.0870 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0830 (3.01) | 0.0850 (23.4) | 0.0910 (5.00) | 0.108 (20.1) | 0.108 (20.1)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 2 | 2 | 3
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  | 0.144 (21.7) |  | 0.0490 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0620 (33.9) | 0.0860 (2.45) | 0.0840 (63.1) | 0.0810 (45.1)
  Total Ab of ADCT-301: Cycle 1 |  | 0.162 (34.6) | 0.0870 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0830 (3.01) | 0.101 (11.7) | 0.0910 (5.00) | 0.119 (31.2) | 0.108 (20.1)
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 2 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  | 0.103 (27.2) |  | 0.0490 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0770 (17.1) | 0.123 (50.2) | 0.0840 (63.1) | 0.0760 (59.1)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  SG3199 Free Warhead of ADCT-301: Cycle 1 |  |  |  |  |  | 0.310 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.379 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.164 (36.1)
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  SG3199 Free Warhead of ADCT-301: Cycle 2 |  |  |  |  |  | 0.228 (12.8) |  | 0.309 (NA) — Standard deviation could not be determined as only one participant had evaluable data.

12. Secondary Outcome: Time to Reach the Maximum Observed Serum Concentration (Tmax) for ADCT-301 for the QW Dosing Schedule
Description: Tmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 5 | 2
days
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1 | 0.0680 (19.9) | 0.119 (173)
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2 | 0.0370 (50.4) | 0.0240 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1 Week 1 | 0.117 (185) | 0.0590 (18.1)
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  Total Ab of ADCT-301: Cycle 1 Week 2 | 0.0370 (50.4) | 0.0240 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ADCT-301 for the Q3W Dosing Schedule
Description: AUClast for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 2 | 1 | 3 | 3 | 3 | 3 | 4
day*μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  | 19.0 (681) | 109 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 34.9 (363) | 317 (43.3) | 897 (67.5) | 1198 (82.1) | 381 (126)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 2 | 2 | 3
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  | 19.1 (7.42) |  | 30.4 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 231 (1225) | 114 (332) | 1063 (135) | 360 (180)
  Total Ab of ADCT-301: Cycle 1 |  | 36.3 (245) | 132 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 46.4 (353) | 590 (40.6) | 1144 (66.7) | 1577 (69.6) | 394 (174)
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3 | 2 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  | 22.6 (23.9) |  | 22.6 (77.7) | 348 (1389) | 127 (452) | 1427 (180) | 436 (178)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  SG3199 Free Warhead of ADCT-301: Cycle 1 |  |  |  |  |  | 0.00500 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0120 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0500 (81.2)
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  SG3199 Free Warhead of ADCT-301: Cycle 2 |  |  |  |  |  | 0.00600 (110) |  | 0.01540 (NA) — Standard deviation could not be determined as only one participant had evaluable data.

14. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ADCT-301 for the QW Dosing Schedule
Description: AUClast for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 5 | 2
day*μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1 | 331 (114) | 113 (86.8)
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2 | 378 (103) | 2319 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1 Week 1 | 476 (116) | 152 (103)
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 4 | 1
  Total Ab of ADCT-301: Cycle 1 Week 2 | 584 (86.8) | 3099 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the End of the Dosing Interval (AUCtau) for ADCT-301 for the Q3W Dosing Schedule
Description: AUCtau for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
day*μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  |  |  |  | 1061 (72.3) | 186 (240) | 1248 (114) | 826 (151)
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  |  |  |  | 1700 (89.6) | 60.2 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1751 (146) | 622 (167)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the End of the Dosing Interval (AUCtau) for ADCT-301 for the QW Dosing Schedule
Description: AUCtau for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: The analysis was planned, but the data was not collected as study was terminated prematurely.
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) for ADCT-301 for the Q3W Dosing Schedule
Description: AUCinf for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
day*μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  |  |  |  |  |  | 2846 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 440 (139)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Total Ab of ADCT-301: Cycle 1 |  |  |  |  | 667 (56.3) | 1631 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 3434 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1019 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) for ADCT-301 for the QW Dosing Schedule
Description: AUCinf for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 1 | 0
day*μg/L
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  Total Ab of ADCT-301: Cycle 1 Week 1 | 366 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Accumulation Index (AI) for ADCT-301 for the Q3W Dosing Schedule
Description: AI for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort. AI is the ratio of area under the serum concentration-time curve (AUC) from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
ratio
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  |  |  |  | 1.00 (0.373) | 1.00 (0) | 1.00 (0.0434) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  |  |  |  | 1.00 (0.416) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.00 (0.113) | 1.00 (0.000222)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Accumulation Index (AI) for ADCT-301 for the QW Dosing Schedule
Description: AI for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort. AI is the ratio of area under the serum concentration-time curve (AUC) from 0 to 7 days divided by AUC from 7 to 14 days for Cycle 1.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 4 | 1
ratio
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 3 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2 | 1.13 (9.77) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  Total Ab of ADCT-301: Cycle 1 Week 2 | 1.12 (14.3) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Volume of Distribution at Steady-state (Vss) for ADCT-301 for the Q3W Dosing Schedule
Description: Vss for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
liters
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  |  |  |  |  |  | 4.27 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 7.34 (120)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  |  |  |  | 6.46 (13.9) | 7.58 (168) | 5.94 (25.7) | 5.29 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Total Ab of ADCT-301: Cycle 1 |  |  |  |  | 5.69 (28.9) | 7.04 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 4.54 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 3.88 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  |  |  |  | 5.74 (2.99) |  | 6.22 (43.3) | 7.83 (37.1)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Volume of Distribution at Steady-state (Vss) for ADCT-301 for the QW Dosing Schedule
Description: Vss for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 1 | 0
liters
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  Total Ab of ADCT-301: Cycle 1 Week 1 | 6.07 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Mean Residence Time (MRT) for ADCT-301 for the Q3W Dosing Schedule
Description: MRT analysis was planned for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Mean Residence Time (MRT) for ADCT-301 for the QW Dosing Schedule
Description: MRT analysis was planned for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Terminal Elimination Phase Rate Constant (λz) for ADCT-301 for the Q3W Dosing Schedule
Description: λz analysis was planned for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Terminal Elimination Phase Rate Constant (λz) for ADCT-301 for the QW Dosing Schedule
Description: λz analysis was planned for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Apparent Terminal Phase Elimination Half-life (Thalf) for ADCT-301 for the Q3W Dosing Schedule
Description: Thalf for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
days
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  |  |  |  |  |  | 2.28 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.446 (45.6)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  |  |  |  | 1.80 (67.7) | 0.379 (63.9) | 1.36 (56.0) | 1.02 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Total Ab of ADCT-301: Cycle 1 |  |  |  |  | 0.995 (45.8) | 2.28 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 2.18 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.587 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  |  |  |  | 1.96 (55.8) |  | 1.57 (55.5) | 0.451 (111)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Apparent Terminal Phase Elimination Half-life (Thalf) for ADCT-301 for the QW Dosing Schedule
Description: Thalf for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 1 | 0
days
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  Total Ab of ADCT-301: Cycle 1 Week 1 | 0.719 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Clearance (CL) for ADCT-301 for the Q3W Dosing Schedule
Description: CL for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for Q3W cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
L/day
  PBD-conjugated Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 1 |  |  |  |  |  |  | 1.67 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 12.5 (237)
  PBD-conjugated Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
  PBD-conjugated Ab of ADCT-301: Cycle 2 |  |  |  |  | 2.68 (40.6) | 14.5 (423) | 3.28 (84.1) | 8.20 (163)
  Total Ab of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Total Ab of ADCT-301: Cycle 1 |  |  |  |  | 4.22 (86.9) | 2.21 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.75 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 5.36 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
  Total Ab of ADCT-301: Cycle 2 |  |  |  |  | 2.12 (54.5) |  | 2.96 (109) | 12.6 (151)
  SG3199 Free Warhead of ADCT-301: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Clearance (CL) for ADCT-301 for the QW Dosing Schedule
Description: CL for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for QW cohort.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
Number analyzed (Participants) | 1 | 0
L/day
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  PBD-conjugated Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  Total Ab of ADCT-301: Cycle 1 Week 1 | 6.59 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |
  Total Ab of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 1: number analyzed (Participants) | 0 | 0
  SG3199 Free Warhead of ADCT-301: Cycle 1 Week 2: number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Number of Participants With Anti-drug Antibody Response (Against ADCT-301)
Description: Blood serum samples were collected and analysed to determine the presence or absence of ADA. Results were pooled for Part 1 participants as specified in the protocol.
Time Frame: Day 1 to the end of Cycle 2 (6 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: ADCT-301 Dose Escalation: Weekly administration: Participants received an IV infusion of ADCT-301, on Days 1, 8, and 15 of each 3-week (21-day) cycle.
  3-week administration: Participants received an IV infusion of ADCT-301, on Day 1 of each 3-week (21-day) cycle.
Arm/Group | Part 1: ADCT-301 Dose Escalation
Number analyzed (Participants) | 34
Participants | 2

ADVERSE EVENTS:
Time Frame: Day 1 to a maximum of 24 weeks (+ 30 days)
Arm/Group | Cohort 1: 3 μg/kg Q3W | Cohort 2: 6 μg/kg Q3W | Cohort 3: 12 μg/kg Q3W | Cohort 4: 22 μg/kg Q3W | Cohort 5: 32 μg/kg Q3W | Cohort 6: 52 μg/kg Q3W | Cohort 7: 72 μg/kg Q3W | Cohort 8: 92 μg/kg Q3W | Cohort 9: 30 μg/kg QW | Cohort 10: 37.5 μg/kg QW
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 2/3 | 2/3 | 2/3 | 1/4 | 5/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 2/3 | 3/3 | 1/3 | 2/3 | 2/3 | 2/4 | 5/6 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 3 μg/kg Q3W (N=4) | Cohort 2: 6 μg/kg Q3W (N=3) | Cohort 3: 12 μg/kg Q3W (N=3) | Cohort 4: 22 μg/kg Q3W (N=3) | Cohort 5: 32 μg/kg Q3W (N=3) | Cohort 6: 52 μg/kg Q3W (N=3) | Cohort 7: 72 μg/kg Q3W (N=3) | Cohort 8: 92 μg/kg Q3W (N=4) | Cohort 9: 30 μg/kg QW (N=6) | Cohort 10: 37.5 μg/kg QW (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Streptococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 3 μg/kg Q3W (N=4) | Cohort 2: 6 μg/kg Q3W (N=3) | Cohort 3: 12 μg/kg Q3W (N=3) | Cohort 4: 22 μg/kg Q3W (N=3) | Cohort 5: 32 μg/kg Q3W (N=3) | Cohort 6: 52 μg/kg Q3W (N=3) | Cohort 7: 72 μg/kg Q3W (N=3) | Cohort 8: 92 μg/kg Q3W (N=4) | Cohort 9: 30 μg/kg QW (N=6) | Cohort 10: 37.5 μg/kg QW (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pupillary Reflex Impaired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Mucosa Haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue Coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Graft versus Host Disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Anorectal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Electrocardiogram QT Prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcus Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin I Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Capillary Leak Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Only a small number of participants were analyzed as the study was early terminated due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT02588092/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02588092/SAP_001.pdf